CLINICAL TRIAL: NCT04850651
Title: A Single-centre, Open, Single-dose, Self-control Study to Investigate the Effect of Fluconazole on the Pharmacokinetics of Pyrotinib in Healthy Chinese Adult Subjects.
Brief Title: Effect of Fluconazole on the Pharmacokinetics of Pyrotinib in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HR-BLTN-DDI-06
Record Dates: First submitted 2021-04-19; First posted 2021-04-20 (Actual); Last update posted 2021-10-22 (Actual); Status verified 2021-10

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Intervention Model Description: Pyrotinib alone and then combination with fluconazole
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pyrotinib/Fluconazole (Experimental): Durg: Pyrotinib Durg: Pyrotinib/Fluconazole Participants received a single oral dose of pyrotinib 80 milligram (mg) on day1 and day9. Participants received a loading dose of fluconazole 400 mg on day6 followed by single dose of fluconazole 200 mg for oral administration from D7 to D18.
  Interventions: Drug: Pyrotinib；Fluconazole

INTERVENTIONS:
Drug: Pyrotinib；Fluconazole — Drug: Pyrotinib Participants received a single oral dose of Pyrotinib tablet on the morning of day1 in treatment period 1.
  Drug: Pyrotinib/Fluconazole In treatment period 2, Participants received a single oral dose of pyrotinib tablet on the morning of day9, and received a loading dose of fluconazole capsule on day6 followed by single dose of fluconazole for oral administration from D7 to D18.

SUMMARY:
The primary objective of the study is to evaluate the effect of fluconazole on pharmacokinetics of pyrotinib tablet for oral administration in healthy Chinese adult subjects. The secondary objective of the study is to compare the safety of pyrotinib alone and co-administered with fluconazole.

ELIGIBILITY:
Inclusion Criteria:

1. Participants has given written informed consent with full understanding of the trial content, process and possible adverse reactions;
2. Ability to complete the study as required by the protocol;
3. Healthy male or female subjects aged 18 to 45 (including 18 and 45) at the date of signing the informed consent;
4. Male body weight ≥ 50 kg, female body weight ≥ 45 kg, and body mass index (BMI) within the range of 19 ~ 26 kg /m2 (including 19 and 26);
5. Willing to take contraception or male subjects who can guarantee not to donate sperm during the trial and within 6 months after the last dose; female subjects with fertility who did not use contraception for at least 2 weeks before dosing;

Exclusion Criteria:

1. Allergic constitution or Allergic to a drug ingredient or component;
2. History of drug use, or drug abuse screening positive;
3. Alcoholic or often drinkers;
4. Left ventricular ejection fraction (LVEF) <50% by echocardiography;
5. A clear medical history of important primary organ diseases such as nervous system, cardiovascular system, urinary system, digestive system, respiratory system, metabolism and musculoskeletal system;
6. Abnormal clinical laboratory tests and clinical significance judged by the investigator or other clinical findings showing the following diseases, including but not limited to gastrointestinal tract, kidney, liver, nerve, blood, endocrine, tumor, lung, immune, mental or cardiovascular and cerebrovascular diseases;
7. Participated in a clinical trial and has received an investigational product within 3 months prior to the first dosing day in the current study;
8. Positive value of HBsAg、HCV-Ab、HIV-Ab、TPPA at screening；
9. Blood loss ≥400mL within 3 months before first dosing;
10. Patients who had a positive blood pregnancy test and were breastfeeding at the time of screening.
11. The investigators determined that other conditions were inappropriate for participation in this clinical trial .

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-16 (Actual); Primary Completion 2021-05-17 (Actual); Study Completion 2021-05-17 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) of Pyrotinib | Pre-dose, and 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 (Combined with Fluconazole), 240 (Combined with Fluconazole) Hours Post-dose
Area Under the Plasma Concentration-Time Curve from Time Zero to Last Measurable Concentration (AUC0-t) of Pyrotinib | Pre-dose, and 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 (Combined with Fluconazole), 240 (Combined with Fluconazole) Hours Post-dose
Area Under the Plasma Concentration-Time Curve from Time Zero to Infinity (AUC0-Inf) of Pyrotinib | Pre-dose, and 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 (Combined with Fluconazole), 240 (Combined with Fluconazole) Hours Post-dose
  AUC0-inf was defined as the area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf).

SECONDARY OUTCOMES:
The Time Take to Reach Cmax (Tmax) of Pyrotinib | Pre-dose, and 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 (Combined with Fluconazole), 240 (Combined with Fluconazole) Hours Post-dose
Elimination Half Life (t1/2) of Pyrotinib | Pre-dose, and 1, 2, 3, 4, 5, 6, 8, 12, 24, 48, 72, 96, 168 (Combined with Fluconazole), 240 (Combined with Fluconazole) Hours Post-dose
  Elimination Half Life (t1/2) was defined as the time required for the concentration or amount of drug in the body to be reduced by one-half.
The Incidence and Severity of Adverse Events (AEs) or Serious Adverse Events (SAEs) in Participants | Baseline up to Day 28

CONTACTS AND LOCATIONS:
Locations (1):
- Jinan Central Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided